CLINICAL TRIAL: NCT02022722
Title: Assessment Of Pain Subsidence And Sexual Function Amelioration Using Either Pelvic Rehabilitation Or Trigger Point Injections
Brief Title: Trigger Point Injections and Pelvic Rehabilitation for the Treatment of Pelvic Floor Myalgia and Sexual Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: Patty Brisben Foundation For Women's Sexual Health (Other)
Responsible Party: Principal Investigator, Mary South, MD, Director of Female Pelvic Medicine & Reconstructive Surgery, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UC IRB Study #: 2013-0677; Patty Brisben Foundation (Other Grant/Funding Number: Patty Brisben Foundation)
Record Dates: First submitted 2013-12-21; First posted 2013-12-30 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Dyspareunia
Keywords: Pelvic Floor Myalgia; Trigger Point Injections; Pelvic Rehabilitation; Dyspareunia
MeSH Terms: conditions — Dyspareunia; Vaginismus | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pelvic Rehabilitation (Active Comparator): Pelvic Rehabilitation will be conduction on weekly basis for a total of 6 weeks
  Interventions: Procedure: Pelvic Rehabilitation
- Trigger Point Injections (Active Comparator): Trigger point injections will be administered on weekly basis for a total of 6 weeks
  Interventions: Drug: Trigger Point Injections Triamcinolone Acetonide, Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Trigger Point Injections Triamcinolone Acetonide, Bupivacaine Hydrochloride — The mixture is injected into the levator muscles, with half the volume on each side of the pelvic musculature.
  Other Names: Triamcinolone Acetonide-Total dose of 40mg, Volume 2 ml; Bupivacaine Hydrochloride-Strength 0.5%, Volume 18ml
  Arms: Trigger Point Injections
Procedure: Pelvic Rehabilitation — Pelvic floor massage will be performed on a weekly basis by a licensed physiotherapist specialized in pelvic floor pelvic therapy
  Other Names: Pelvic floor massage
  Arms: Pelvic Rehabilitation

SUMMARY:
The purpose of this study is to evaluate which treatment option for pelvic floor pain allows for improved sexual function.

DETAILED DESCRIPTION:
Pelvic floor pain may be treated with trigger point injections with medications (steroids and local anesthetics) that are FDA approved for injection into muscles. The alternative is a noninvasive treatment option using pelvic rehabilitation which involves vaginal muscle massage. Both treatment options have been used and reported; however, rapidity of improvement and return to normal sexual function have not been assessed. This study assigns patients to either treatment option randomly and the sexual function is assessed based on standardized sexual function questionnaires as well as pain ratings.

ELIGIBILITY:
Inclusion Criteria:

* pelvic pain
* pelvic floor myalgia
* dyspareunia
* female
* age > 18 years

Exclusion Criteria:

* interstitial cystitis
* vaginal lesions / ulcerations
* prior trigger point injections in the past 6 months
* prior pelvic rehabilitation in the past 6 months
* laparoscopically documented endometriosis / pelvic adhesions or adhesive disease
* documented pelvic inflammatory disease identified within the past 6 months
* documented sexually transmitted disease within the past 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-04 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Change in rating of pain from baseline until the end of the study according to the Iowa Pain Scale | Baseline, Week 10
  Patients will be asked to rate their current pain prior to initiation of the treatment at the visits, at the start of the study and after the completion of the study, using the 10 point Iowa Pain scale.

SECONDARY OUTCOMES:
Change in sexual function between visit 1 and visit 10 | Baseline, Week 10
  Change in sexual function based on the female sexual function index (19 questions, one final score, maximum score of 36) where the patients fill a questionnaire prior to the first treatment session and after the completion of the treatment at week 10.

CONTACTS AND LOCATIONS:
Overall Officials: Mary South, MD, Principal Investigator — University of Cincinnati
Locations (1):
- Division of Urogynecology, University of Cincinnati Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Mathias SD, Kuppermann M, Liberman RF, Lipschutz RC, Steege JF. Chronic pelvic pain: prevalence, health-related quality of life, and economic correlates. Obstet Gynecol. 1996 Mar;87(3):321-7. doi: 10.1016/0029-7844(95)00458-0. PMID 8598948
- [Result] Rao SS, Paulson J, Mata M, Zimmerman B. Clinical trial: effects of botulinum toxin on Levator ani syndrome--a double-blind, placebo-controlled study. Aliment Pharmacol Ther. 2009 May 1;29(9):985-91. doi: 10.1111/j.1365-2036.2009.03964.x. Epub 2009 Feb 13. PMID 19222415
- [Result] Langford CF, Udvari Nagy S, Ghoniem GM. Levator ani trigger point injections: An underutilized treatment for chronic pelvic pain. Neurourol Urodyn. 2007;26(1):59-62. doi: 10.1002/nau.20393. PMID 17195176
- [Result] Jarvis SK, Abbott JA, Lenart MB, Steensma A, Vancaillie TG. Pilot study of botulinum toxin type A in the treatment of chronic pelvic pain associated with spasm of the levator ani muscles. Aust N Z J Obstet Gynaecol. 2004 Feb;44(1):46-50. doi: 10.1111/j.1479-828X.2004.00163.x. PMID 15089868